CLINICAL TRIAL: NCT04811521
Title: Patient-centered Treatment of Anxiety After Low-Risk Chest Pain in the Emergency Room
Acronym: PACER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Paul Musey, Director of Research, Indiana University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10296
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Generalized Anxiety Disorder; Chest Pain; Panic
MeSH Terms: conditions — Generalized Anxiety Disorder; Chest Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primary care follow-up (Active Comparator): Enhanced primary care coordination
  Interventions: Behavioral: Primary care follow-up
- Online Cognitive Behavioral Therapy (Active Comparator): Online Self-Administered Anxiety Management Program plus Peer Support Guidance
  Interventions: Behavioral: Online Self-Administered Anxiety Management Program plus Peer Support Guidance
- Therapist-Administered Cognitive Behavioral Therapy (Active Comparator): Telehealth 8 one-hour sessions over the course of 8 to 10 weeks
  Interventions: Behavioral: Therapist-Administered Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Primary care follow-up — Those randomized to primary care and enhanced primary care coordination will receive the minimal intensity treatment that includes: (1) assistance in identifying a primary care provider for participants who do not have one, (2) sharing results of diagnostic testing (including anxiety screening) with the primary care provider (results sent via EMR note, mailed letter, or delivered by participant at appointment); and (3) an educational brochure on anxiety and treatment.
  Arms: Primary care follow-up
Behavioral: Online Self-Administered Anxiety Management Program plus Peer Support Guidance — Individuals randomized to the online Cognitive Behavioral Therapy (CBT) + peer support guidance arm will receive access to six online, evidence-based CBT modules in the This Way Up Generalized Anxiety Course to be completed weekly or bi-monthly. Individuals who screen positive on the PHQ panic measure will complete 2 additional panic-specific homework assignments applying exposure therapy to panic (in addition to Generalized Anxiety Disorder) experiences aligned with content from the This Way Up Panic Course.
  Arms: Online Cognitive Behavioral Therapy
Behavioral: Therapist-Administered Cognitive Behavioral Therapy — Individuals randomized to therapist-led CBT via telehealth will receive 8 one-hour sessions over the course of 8 to 10 weeks via telehealth (HIPAA compliant software such as Zoom Health or AmWell) or telephone. Therapists will be master's-degreed or eligible clinicians trained in CBT by our study psychologist. Therapists will follow a manualized protocol for delivering CBT for anxiety, specifically, with a primary focus on anxiety and worry management. Individuals who screen positive on the PHQ panic measure will have training in exposure therapy added to CBT. Although many CBT trials have a standard length of 12 sessions, brief CBT lasting 4-8 sessions is equally efficacious.
  Arms: Therapist-Administered Cognitive Behavioral Therapy

SUMMARY:
The goal of this research is to compare the benefits and risks of three anxiety treatments that are pragmatic, graduated in the level of resource intensity, and have demonstrated efficacy and feasibility for real world adoption.

DETAILED DESCRIPTION:
The goal of this research is to compare the benefits and risks of three anxiety treatments that are pragmatic, graduated in the level of resource intensity, and have demonstrated efficacy and feasibility for real world adoption. Low-risk (non-cardiac) chest pain patients with anxiety will be recruited to participate in the study using the SBIRT (screening, brief intervention, and referral to treatment) model and enrolled participants will be randomly assigned to one of three treatment arms: 1) referral to primary care with enhanced care coordinated (low intensity); 2) online CBT with support from a certified peer recovery specialist (medium intensity); and 3) therapist-led CBT via tele-health (high intensity). We expect improved symptoms and functional capacity, reduced ED return visits, and heterogenous treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult emergency department (ED) patients (≥18yoa) presenting to the ED
* Within 1 week of ED presentation if discharged at time of screening.
* Chief complaint of chest pain or similar chief complaint leading to a standard of care diagnostic protocol to rule out possible acute coronary syndrome.
* HEART Score of 0-3 indicating Major Adverse Cardiac Events (MACE) risk equivalent to ≤2%
* "Functionally" low risk status - (moderate HEART score of 4-6) plus diagnostic protocol evaluation with at least two serial normal troponins spaced at least six hours apart with or without cardiovascular stress testing in the observation unit.
* Moderate to severe anxiety as defined by a GAD-7 score ≥ 8 or a PHQ panic screener score ≥ 2
* Expected to be discharged from the ED or only undergo observation <24 hours.

Exclusion Criteria:

* > 1 week from ED discharge
* Traumatic reason for chest pain
* Those admitted to the hospital (inpatient status) as part of their ED presentation (those placed in the observation unit for planned observation less than <24 hours are eligible)
* Active psychosis or behavioral issues requiring psychiatric monitoring or consultation of psychiatry for psychosis, schizophrenia, or suicidal ideation
* Hemodynamic instability as assessed by the treating provider
* Issues likely to affect follow up, including prisoners and homelessness
* Inability to understand and speak English to participate in telehealth therapy sessions and peer support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-08-17 (Estimated); Study Completion 2025-08-17 (Estimated)

PRIMARY OUTCOMES:
Anxiety Symptoms | 3 months after enrollment
  General Anxiety Disorder-7 scale score adjusted for baseline. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Anxiety Symptoms | 6 months after enrollment
  General Anxiety Disorder-7 scale score adjusted for baseline. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Anxiety Symptoms | 9 months after enrollment
  General Anxiety Disorder-7 scale score adjusted for baseline. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
Anxiety Symptoms | 12 months after enrollment
  General Anxiety Disorder-7 scale score adjusted for baseline. 0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety

SECONDARY OUTCOMES:
Panic Symptoms | 3 months after enrollment
  PHQ Panic Screener adjusted for baseline
Panic Symptoms | 6 months after enrollment
  PHQ Panic Screener adjusted for baseline
Panic Symptoms | 9 months after enrollment
  PHQ Panic Screener adjusted for baseline
Panic Symptoms | 12 months after enrollment
  PHQ Panic Screener adjusted for baseline
Chest Pain | 3 months after enrollment
  Chest pain frequency as adjusted for baseline
Chest Pain | 6 months after enrollment
  Chest pain frequency as adjusted for baseline
Chest Pain | 9 months after enrollment
  Chest pain frequency as adjusted for baseline
Chest Pain | 12 months after enrollment
  Chest pain frequency as adjusted for baseline
Physical Symptoms | 3 months after enrollment
  PHQ-15 total score as adjusted for baseline
Physical Symptoms | 6 months after enrollment
  PHQ-15 total score as adjusted for baseline
Physical Symptoms | 9 months after enrollment
  PHQ-15 total score as adjusted for baseline
Physical Symptoms | 12 months after enrollment
  PHQ-15 total score as adjusted for baseline
Depression symptoms | 3 months after enrollment
  PHQ-8 total score as adjusted for baseline
Depression symptoms | 6 months after enrollment
  PHQ-8 total score as adjusted for baseline
Depression symptoms | 9 months after enrollment
  PHQ-8 total score as adjusted for baseline
Depression symptoms | 12 months after enrollment
  PHQ-8 total score as adjusted for baseline
Work/family/social functioning | 3 months after enrollment
  Sheehan Disability scale as adjusted for baseline
Work/family/social functioning | 6 months after enrollment
  Sheehan Disability scale as adjusted for baseline
Work/family/social functioning | 9 months after enrollment
  Sheehan Disability scale as adjusted for baseline
Work/family/social functioning | 12 months after enrollment
  Sheehan Disability scale as adjusted for baseline
Global Anxiety Change | 3 months after enrollment
  Patient-rated global anxiety change since enrollment
Global Anxiety Change | 6 months after enrollment
  Patient-rated global anxiety change since enrollment
Global Anxiety Change | 9 months after enrollment
  Patient-rated global anxiety change since enrollment
Global Anxiety Change | 12 months after enrollment
  Patient-rated global anxiety change since enrollment
ED Utilization | 12 months prior to enrollment
  Number of return visits to ED
ED Utilization | 3 months after enrollment
  Number of return visits to ED
ED Utilization | 6 months after enrollment
  Number of return visits to ED
ED Utilization | 9 months after enrollment
  Number of return visits to ED
ED Utilization | 12 months after enrollment
  Number of return visits to ED
Adverse Cardiac Events | 3 months after enrollment
  Number of major adverse cardiac events (death, myocardial infarction, revascularization)
Adverse Cardiac Events | 6 months after enrollment
  Number of major adverse cardiac events (death, myocardial infarction, revascularization)
Adverse Cardiac Events | 9 months after enrollment
  Number of major adverse cardiac events (death, myocardial infarction, revascularization)
Adverse Cardiac Events | 12 months after enrollment
  Number of major adverse cardiac events (death, myocardial infarction, revascularization)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Musey, MD, Principal Investigator — Indiana University
Locations (5):
- United States (5):
  - Indiana University Health West Hospital, Avon, Indiana
  - Indiana University Health North Hospital, Carmel, Indiana
  - Indiana University Health Saxony Hospital, Fishers, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University Health Ball Memorial Hosptial, Muncie, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rui P, Kang K. National Hospital Ambulatory Medical Care Survey: 2015 Emergency Department Summary Tables. CDC, US Centers for Disease Control and Prevention; 2015:34.
- [Background] Kline JA, Shapiro NI, Jones AE, Hernandez J, Hogg MM, Troyer J, Nelson RD. Outcomes and radiation exposure of emergency department patients with chest pain and shortness of breath and ultralow pretest probability: a multicenter study. Ann Emerg Med. 2014 Mar;63(3):281-8. doi: 10.1016/j.annemergmed.2013.09.009. Epub 2013 Oct 10. PMID 24120629
- [Background] Eslick GD, Talley NJ. Natural history and predictors of outcome for non-cardiac chest pain: a prospective 4-year cohort study. Neurogastroenterol Motil. 2008 Sep;20(9):989-97. doi: 10.1111/j.1365-2982.2008.01133.x. Epub 2008 May 6. PMID 18466221
- [Background] Musey PI Jr, Patel R, Fry C, Jimenez G, Koene R, Kline JA. Anxiety Associated With Increased Risk for Emergency Department Recidivism in Patients With Low-Risk Chest Pain. Am J Cardiol. 2018 Oct 1;122(7):1133-1141. doi: 10.1016/j.amjcard.2018.06.044. Epub 2018 Jul 5. PMID 30086878
- [Background] Webster R, Norman P, Goodacre S, Thompson AR, McEachan RR. Illness representations, psychological distress and non-cardiac chest pain in patients attending an emergency department. Psychol Health. 2014;29(11):1265-82. doi: 10.1080/08870446.2014.923885. Epub 2014 Jun 18. PMID 24831735
- [Background] Foldes-Busque G, Marchand A, Chauny JM, Poitras J, Diodati J, Denis I, Lessard MJ, Pelland ME, Fleet R. Unexplained chest pain in the ED: could it be panic? Am J Emerg Med. 2011 Sep;29(7):743-51. doi: 10.1016/j.ajem.2010.02.021. Epub 2010 May 1. PMID 20825891
- [Background] Demiryoguran NS, Karcioglu O, Topacoglu H, Kiyan S, Ozbay D, Onur E, Korkmaz T, Demir OF. Anxiety disorder in patients with non-specific chest pain in the emergency setting. Emerg Med J. 2006 Feb;23(2):99-102. doi: 10.1136/emj.2005.025163. PMID 16439735
- [Background] Eken C, Oktay C, Bacanli A, Gulen B, Koparan C, Ugras SS, Cete Y. Anxiety and depressive disorders in patients presenting with chest pain to the emergency department: a comparison between cardiac and non-cardiac origin. J Emerg Med. 2010 Aug;39(2):144-50. doi: 10.1016/j.jemermed.2007.11.087. Epub 2008 Aug 23. PMID 18722737
- [Background] Aikens JE, Michael E, Levin T, Myers TC, Lowry E, McCracken LM. Cardiac exposure history as a determinant of symptoms and emergency department utilization in noncardiac chest pain patients. J Behav Med. 1999 Dec;22(6):605-17. doi: 10.1023/a:1018745813664. PMID 10650539
- [Background] Hunot V, Churchill R, Silva de Lima M, Teixeira V. Psychological therapies for generalised anxiety disorder. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD001848. doi: 10.1002/14651858.CD001848.pub4. PMID 17253466
- [Background] Kisely SR, Campbell LA, Yelland MJ, Paydar A. Psychological interventions for symptomatic management of non-specific chest pain in patients with normal coronary anatomy. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD004101. doi: 10.1002/14651858.CD004101.pub4. PMID 22696339
- [Background] Nault Connors JD, Prittie A, Musey PI. Why an Algorithmic "Rule-Out MI" Order Set Is Necessary But Not Sufficient Care for Chest Pain in the Emergency Department Setting. J Patient Exp. 2020 Oct;7(5):685-687. doi: 10.1177/2374373519881279. Epub 2019 Oct 15. No abstract available. PMID 33294601
- [Background] Napoli AM, Baird J, Tran S, Wang J. Low Adverse Event Rates But High Emergency Department Utilization in Chest Pain Patients Treated in an Emergency Department Observation Unit. Crit Pathw Cardiol. 2017 Mar;16(1):15-21. doi: 10.1097/HPC.0000000000000099. PMID 28195938
- [Background] Backus BE, Six AJ, Kelder JC, Bosschaert MA, Mast EG, Mosterd A, Veldkamp RF, Wardeh AJ, Tio R, Braam R, Monnink SH, van Tooren R, Mast TP, van den Akker F, Cramer MJ, Poldervaart JM, Hoes AW, Doevendans PA. A prospective validation of the HEART score for chest pain patients at the emergency department. Int J Cardiol. 2013 Oct 3;168(3):2153-8. doi: 10.1016/j.ijcard.2013.01.255. Epub 2013 Mar 7. PMID 23465250
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Craske MG, Stein MB, Sullivan G, Sherbourne C, Bystritsky A, Rose RD, Lang AJ, Welch S, Campbell-Sills L, Golinelli D, Roy-Byrne P. Disorder-specific impact of coordinated anxiety learning and management treatment for anxiety disorders in primary care. Arch Gen Psychiatry. 2011 Apr;68(4):378-88. doi: 10.1001/archgenpsychiatry.2011.25. PMID 21464362
- [Background] Rodriguez BF, Weisberg RB, Pagano ME, Machan JT, Culpepper L, Keller MB. Frequency and patterns of psychiatric comorbidity in a sample of primary care patients with anxiety disorders. Compr Psychiatry. 2004 Mar-Apr;45(2):129-37. doi: 10.1016/j.comppsych.2003.09.005. PMID 14999664
- [Background] Lowe B, Grafe K, Zipfel S, Spitzer RL, Herrmann-Lingen C, Witte S, Herzog W. Detecting panic disorder in medical and psychosomatic outpatients: comparative validation of the Hospital Anxiety and Depression Scale, the Patient Health Questionnaire, a screening question, and physicians' diagnosis. J Psychosom Res. 2003 Dec;55(6):515-9. doi: 10.1016/s0022-3999(03)00072-2. PMID 14642981
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Perini S, Titov N, Andrews G. Clinician-assisted Internet-based treatment is effective for depression: randomized controlled trial. Aust N Z J Psychiatry. 2009 Jun;43(6):571-8. doi: 10.1080/00048670902873722. PMID 19440890
- [Background] Mewton L, Wong N, Andrews G. The effectiveness of internet cognitive behavioural therapy for generalized anxiety disorder in clinical practice. Depress Anxiety. 2012 Oct;29(10):843-9. doi: 10.1002/da.21995. Epub 2012 Sep 4. PMID 22949296
- [Background] Dugas MJ, Robichaud M. Cognitive-Behavioral Treatment for Generalized Anxiety Disorder: From Science to Practice. New York. : Routledge; 2007.
- [Background] Cape J, Whittington C, Buszewicz M, Wallace P, Underwood L. Brief psychological therapies for anxiety and depression in primary care: meta-analysis and meta-regression. BMC Med. 2010 Jun 25;8:38. doi: 10.1186/1741-7015-8-38. PMID 20579335
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Mitchell AJ, Yadegarfar M, Gill J, Stubbs B. Case finding and screening clinical utility of the Patient Health Questionnaire (PHQ-9 and PHQ-2) for depression in primary care: a diagnostic meta-analysis of 40 studies. BJPsych Open. 2016 Mar 9;2(2):127-138. doi: 10.1192/bjpo.bp.115.001685. eCollection 2016 Mar. PMID 27703765
- [Background] Zijlema WL, Stolk RP, Lowe B, Rief W; BioSHaRE; White PD, Rosmalen JG. How to assess common somatic symptoms in large-scale studies: a systematic review of questionnaires. J Psychosom Res. 2013 Jun;74(6):459-68. doi: 10.1016/j.jpsychores.2013.03.093. Epub 2013 Apr 24. PMID 23731742
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Leon AC, Olfson M, Portera L, Farber L, Sheehan DV. Assessing psychiatric impairment in primary care with the Sheehan Disability Scale. Int J Psychiatry Med. 1997;27(2):93-105. doi: 10.2190/T8EM-C8YH-373N-1UWD. PMID 9565717
- [Background] Leon AC, Shear MK, Portera L, Klerman GL. Assessing impairment in patients with panic disorder: the Sheehan Disability Scale. Soc Psychiatry Psychiatr Epidemiol. 1992 Mar;27(2):78-82. doi: 10.1007/BF00788510. PMID 1594977
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Kroenke K, Krebs E, Wu J, Bair MJ, Damush T, Chumbler N, York T, Weitlauf S, McCalley S, Evans E, Barnd J, Yu Z. Stepped Care to Optimize Pain care Effectiveness (SCOPE) trial study design and sample characteristics. Contemp Clin Trials. 2013 Mar;34(2):270-81. doi: 10.1016/j.cct.2012.11.008. Epub 2012 Dec 8. PMID 23228858
- [Background] Krebs EE, Gravely A, Nugent S, Jensen AC, DeRonne B, Goldsmith ES, Kroenke K, Bair MJ, Noorbaloochi S. Effect of Opioid vs Nonopioid Medications on Pain-Related Function in Patients With Chronic Back Pain or Hip or Knee Osteoarthritis Pain: The SPACE Randomized Clinical Trial. JAMA. 2018 Mar 6;319(9):872-882. doi: 10.1001/jama.2018.0899. PMID 29509867
- [Background] Kroenke K, Evans E, Weitlauf S, McCalley S, Porter B, Williams T, Baye F, Lourens SG, Matthias MS, Bair MJ. Comprehensive vs. Assisted Management of Mood and Pain Symptoms (CAMMPS) trial: Study design and sample characteristics. Contemp Clin Trials. 2018 Jan;64:179-187. doi: 10.1016/j.cct.2017.10.006. Epub 2017 Oct 12. PMID 29031492
- [Background] Prins A, Ouimette P, Kimerling R. The primary care PTSD screen (PC-PTSD): development and operating characteristics. Primary Care Psychiatry 2003;9:9-14.
- [Background] Reichheld FF. The one number you need to grow. Harv Bus Rev. 2003 Dec;81(12):46-54, 124. PMID 14712543
- [Background] Bushey MA, Kroenke K, Weiner J, Porter B, Evans E, Baye F, Lourens S, Weitlauf S. Telecare management of pain and mood symptoms: Adherence, utility, and patient satisfaction. J Telemed Telecare. 2020 Dec;26(10):619-626. doi: 10.1177/1357633X19856156. Epub 2019 Jun 20. PMID 31221047
- [Background] Schwarzer R, Born A. Optimistic self-beliefs: Assessment of general perceived self-efficacy in thirteen cultures. World Psychology 1997;3:177-90.
- [Background] Eich HS, Kriston L, Schramm E, Bailer J. The German version of the helping alliance questionnaire: psychometric properties in patients with persistent depressive disorder. BMC Psychiatry. 2018 Apr 23;18(1):107. doi: 10.1186/s12888-018-1697-8. PMID 29685124
- [Background] Granner ML, Sharpe PA. Evaluating community coalition characteristics and functioning: a summary of measurement tools. Health Educ Res. 2004 Oct;19(5):514-32. doi: 10.1093/her/cyg056. Epub 2004 May 17. PMID 15150134
- [Background] Butterfoss FD, Goodman RM, Wandersman A. Community coalitions for prevention and health promotion. Health Educ Res. 1993 Sep;8(3):315-30. doi: 10.1093/her/8.3.315. No abstract available. PMID 10146473
- [Background] Kroenke K, Baye F, Lourens SG, Evans E, Weitlauf S, McCalley S, Porter B, Matthias MS, Bair MJ. Automated Self-management (ASM) vs. ASM-Enhanced Collaborative Care for Chronic Pain and Mood Symptoms: the CAMMPS Randomized Clinical Trial. J Gen Intern Med. 2019 Sep;34(9):1806-1814. doi: 10.1007/s11606-019-05121-4. Epub 2019 Jun 21. PMID 31228055
- [Background] Dube P, Kurt K, Bair MJ, Theobald D, Williams LS. The p4 screener: evaluation of a brief measure for assessing potential suicide risk in 2 randomized effectiveness trials of primary care and oncology patients. Prim Care Companion J Clin Psychiatry. 2010;12(6):PCC.10m00978. doi: 10.4088/PCC.10m00978blu. PMID 21494337
- [Background] Kroenke K, Krebs EE, Wu J, Yu Z, Chumbler NR, Bair MJ. Telecare collaborative management of chronic pain in primary care: a randomized clinical trial. JAMA. 2014 Jul 16;312(3):240-8. doi: 10.1001/jama.2014.7689. PMID 25027139
- [Background] Muthen LK, Muthen BO. Mplus User's Guide. Eighth Edition. Los Angeles, CA: Muthen & Muthen; 1998-2017.
- [Background] Reichheld FF, Markey R. The Ultimate Question 2.0: How Net Promoter Companies Thrive in a Customer-driven World: Harvard Business Press; 2011.
- [Background] Cohen J. Statistical power analysis for the behavioral sciences. 2nd ed. New York: Academic Press; 1988.
- [Background] Benjamini Y, Hochberg Y. Controlling the false discovery rate: A practical and powerful approach to multiple testing. Journal of the Royal Statistical Society, Series B (Methodological) 1995;57:289-300.
- [Background] Richards DA, Suckling R. Improving access to psychological therapies: phase IV prospective cohort study. Br J Clin Psychol. 2009 Nov;48(Pt 4):377-96. doi: 10.1348/014466509X405178. Epub 2009 Feb 9. PMID 19208291
- [Background] Ali S, Rhodes L, Moreea O, McMillan D, Gilbody S, Leach C, Lucock M, Lutz W, Delgadillo J. How durable is the effect of low intensity CBT for depression and anxiety? Remission and relapse in a longitudinal cohort study. Behav Res Ther. 2017 Jul;94:1-8. doi: 10.1016/j.brat.2017.04.006. Epub 2017 Apr 18. PMID 28437680
- [Derived] He A, Kroenke K, Stump T, Monahan PO, Connors J, Chernyak Y, Musey P. The patient health questionnaire somatization-anxiety-depression scale: Validation of the PHQ-SAD in 4 clinical trials. J Affect Disord. 2026 Apr 1;398:120906. doi: 10.1016/j.jad.2025.120906. Epub 2025 Dec 21. PMID 41436014
- [Derived] Dang L, Kroenke K, Connors J, Stump TE, Monahan PO, Chernyak Y, Holmes E, Hoffman C, Prather K, Musey PI. Psychological Comorbidity in Patients Presenting to the Emergency Department With Low-Risk Chest Pain and Anxiety. Acad Emerg Med. 2026 Jan;33(1):e70113. doi: 10.1111/acem.70113. Epub 2025 Aug 8. PMID 40781746
- [Derived] Connors JN, Kroenke K, Monahan P, Chernyak Y, Pettit K, Hayden J, Montgomery C, Brenner G, Millard M, Holmes E, Musey P. Comparing the effectiveness of existing anxiety treatment options among patients evaluated for chest pain and anxiety in the emergency department setting: Study protocol for the PACER pragmatic randomized comparative effectiveness trial. Contemp Clin Trials. 2023 Jan;124:107020. doi: 10.1016/j.cct.2022.107020. Epub 2022 Nov 21. PMID 36423863